CLINICAL TRIAL: NCT06274125
Title: The Assessment of Kidney Damage Using NGAL Measurements in Patients Undergoing Robotic Radical Prostatectomy
Brief Title: Evaluation of Kidney Damage Using NGAL Measurements
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: AslıDemircioglu1
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Prostatectomy; Neutrophil Gelatinase-Associated Lipocalin; Kidney Function Tests
Keywords: robotic surgery; Neutrophil Gelatinase-Associated Lipocalin; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Preoperative and perioperative blood samples will be taken at the 2nd and 6th hours to determine NGAL values. Blood samples will also be taken for urea, creatinine, and GFR values.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NGAL measurement for evaluating kidney damage in patients undergoing robotic radical prostatectomy.: For the evaluation of kidney damage in patients undergoing robotic radical prostatectomy, blood samples will be collected at preoperative and perioperative 2nd and 6th hours to measure NGAL values.
  Interventions: Procedure: Robotic-Assisted Laparoscopic Radical Prostatectomy

INTERVENTIONS:
Procedure: Robotic-Assisted Laparoscopic Radical Prostatectomy — To evaluate kidney damage in patients undergoing robotic radical prostatectomy, NGAL measurement will be performed.

SUMMARY:
The main objective of this study is to evaluate whether blood NGAL measurement provides superiority over sCr and BUN tests in early diagnosis for assessing renal function in patients undergoing robotic urological surgery.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate whether blood NGAL measurement provides superiority over sCr and BUN tests in early diagnosis for assessing renal function in patients undergoing robotic urological surgery.

The secondary objective of the study is to evaluate the relationship between AKI development and monitored parameters such as age, BMI, comorbidities, ASA, OAB (overactive bladder), mean arterial pressure, intraabdominal pressure, surgical duration, urea and creatinine levels.

After obtaining ethical approval from the Ministry of Health Ankara City Hospital Oncology Operating Room, a total of 55 patients between the ages of 18-80, ASA 1-3, who will undergo general anesthesia under elective conditions will be included in this prospective observational study.

During the preoperative period, patients will be evaluated and provided with written informed consent. Before being taken to the operating room, patients' age, gender, weight, height, body mass index (BMI), comorbidities, regular medication use, ASA classification, hemodynamic values and laboratory values will be recorded in the waiting area. Once in the operating room, patients will be monitored according to the standard working protocol of the anesthesia clinic including non-invasive arterial blood pressure monitoring, 3 or 5-channel ECG and pulse oximetry. Additionally, standard preoperative and postoperative biochemical profiles (including hemogram) and urinary NGAL levels will be measured.

During the perioperative period, routine hemodynamic parameters such as heart rate (HR) (beats per minute), systolic arterial blood pressure (SAB) (mmHg), diastolic arterial blood pressure (DAB) (mmHg), mean arterial blood pressure (OAB)(mmHg), peripheral oxygen saturation(SpO2) as well as postoperative laboratory values will be recorded.

Blood samples for NGAL measurements will be collected at preoperative and perioperative hours 2nd and 6th. Creatinine clearance calculation,hourly urine output; which are commonly used markers to evaluate acute kidney injury(AKI) along with standard laboratory parameters,and other complications related to AKI management ,will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* A total of 55 patients, with ASA scores 1-2-3, aged between 18 and 80 years, will be included in the study conducted at the Robotic Surgery operating room of Ankara City Hospital, Ministry of Health, Turkey.

Exclusion Criteria:

-1. Individuals who do not have the ability to read, understand, or sign the consent form.

2. Individuals with diagnosed renal disease. 3. Patients who do not wish to participate in the study. 4. Patients classified as ASA-3 or higher.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants were selected from male individuals as the evaluation was conducted on patients undergoing prostatectomy.
Study Population: A total of 55 patients, with ASA scores 1-2-3, aged between 18 and 80 years, will be included in the study conducted at the Robotic Surgery operating room of Ankara City Hospital, Ministry of Health, Turkey.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
The main objective of this study is to evaluate whether blood NGAL measurement has superiority over sCr and BUN tests in terms of early diagnosis for assessing kidney function in patients undergoing robotic urologic surgery. | For the evaluation of kidney damage in patients undergoing robotic radical prostatectomy, blood samples will be collected at preoperative and perioperative 2nd and 6th hours to measure NGAL values.

SECONDARY OUTCOMES:
The relationship between demographic parameters such as age, BMI, comorbidities, and ASA classification will be evaluated in relation to the development of AKI. | For the evaluation of kidney damage in patients undergoing robotic radical prostatectomy, blood samples will be collected at preoperative and perioperative 2nd and 6th hours to measure NGAL values.
The evaluation of the relationship between intraabdominal pressure and the development of AKI. | The relationship between intraabdominal pressure monitoring during surgery and NGAL values obtained at 0, 2, and 6 hours.
The relationship between intraoperative mean arterial pressure (MAP) and NGAL (Neutrophil Gelatinase-Associated Lipocalin) values. | The relationship between intraoperative mean arterial pressure monitoring and NGAL values obtained at 0, 2, and 6 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Savran Karadeniz M, Alp Eniste I, Senturk Ciftci H, Usta S, Tefik T, Sanli O, Pembeci K, Tugrul KM. Neutrophil Gelatinase-associated Lipocalin Significantly Correlates with Ischemic Damage in Patients Undergoing Laparoscopic Partial Nephrectomy. Balkan Med J. 2019 Feb 28;36(2):121-128. doi: 10.4274/balkanmedj.galenos.2018.2018.0852. Epub 2018 Nov 12. PMID 30417831
- [Result] Orsolya M, Attila-Zoltan M, Gherman V, Zaharie F, Bolboaca S, Chira C, Bodolea C, Tomuleasa C, Irimie A, Coman I, Ionescu D. The effect of anaesthetic management on neutrophil gelatinase associated lipocalin (NGAL) levels after robotic surgical oncology. J BUON. 2015 Jan-Feb;20(1):317-24. PMID 25778333
- [Result] Buonafine M, Martinez-Martinez E, Jaisser F. More than a simple biomarker: the role of NGAL in cardiovascular and renal diseases. Clin Sci (Lond). 2018 May 8;132(9):909-923. doi: 10.1042/CS20171592. Print 2018 May 16. PMID 29739822
- [Result] Shavit L, Dolgoker I, Ivgi H, Assous M, Slotki I. Neutrophil gelatinase-associated lipocalin as a predictor of complications and mortality in patients undergoing non-cardiac major surgery. Kidney Blood Press Res. 2011;34(2):116-24. doi: 10.1159/000323897. Epub 2011 Feb 11. PMID 21311195
- [Result] Akpinar C, Dogan O, Kubilay E, Gokce MI, Suer E, Gulpinar O, Baltaci S. The evaluation of acute kidney injury due to ischemia by urinary neutrophil gelatinase-induced lipocalin (uNGAL) measurement in patients who underwent partial nephrectomy. Int Urol Nephrol. 2021 Mar;53(3):393-400. doi: 10.1007/s11255-020-02660-2. Epub 2020 Sep 26. PMID 32980930
- [Result] Colamonico O, Cardo G, Ceci E, Scarcia M, Zazzara M, Dassira M, Porreca A, Ludovico GM. The variation of selective uNGAL levels after robot-assisted partial nephrectomy: Early results of a prospective single center study. Arch Ital Urol Androl. 2019 Jul 2;91(2). doi: 10.4081/aiua.2019.2.74. PMID 31266271